CLINICAL TRIAL: NCT05680272
Title: The Effect of Empathic Communication-Based Education on Women's Positive Birth Perception Awareness and Birth Experience
Brief Title: Women's Positive Birth Perception Awareness and Birth Experience
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Emine Aksut Akcay, Lecturer, Kahramanmaras Sutcu Imam University
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: TRKMARAŞ46
Record Dates: First submitted 2022-12-29; First posted 2023-01-11 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Pregnancy Related
Keywords: Pregnancy; Scale; Empathic Communication; Positive Perception of Birth; Midwifery Care

STUDY DESIGN:
Intervention Model Description: education-centered randomized controlled experimental study
Masking Description: In the first stage of the research, it is planned to take a sample of at least 5-10 times the number of items of the scale planned to be developed. The sample size should be at least 200 to reveal the psychometric structure of the scale adequately, 300 and ideally over 500 to reveal the factor structure. In the second phase, it is aimed to reach at least 72 people, 36 in the intervention group and 36 in the control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- extrimental group (Experimental): The experimental group will be given training on empathetic communication and the positive birth perception awareness scale will be applied to the experimental group.
  Interventions: Behavioral: empathic communication-based education
- control group (No Intervention): No intervention will be made in the control group.

INTERVENTIONS:
Behavioral: empathic communication-based education — The study will consist of two stages. The first stage will be methodological in order to develop the Positive Birth Perception Awareness Scale based on Empathic Communication, and the second stage will be a trial model with a pretest-posttest control group in order to determine the effect of the training given to pregnant women based on empathic communication on positive birth perception awareness and birth experience.
  Arms: extrimental group

SUMMARY:
it was aimed to determine the effect of empathic communication-based education on positive birth perception awareness.

DETAILED DESCRIPTION:
Since the existence of humanity, women have not been left alone during pregnancy, childbirth and postpartum period in all societies, but have been supported by their environment. In providing this support, midwives have important responsibilities as the primary responsible health professional . Quality midwifery care given at birth is very important for women to have a positive birth experience The biggest expectations of mothers from midwives in the birth and postpartum period are; it is approaching with empathetic communication such as smiling, therapeutic touch, listening, speaking in a language that the pregnant can understand, making oneself feel good, encouraging, informing, paying attention to privacy. Mothers whose expectations are met in labor; It can have positive obstetric outcomes such as shortening the delivery time, reduction in analgesia and medical intervention applications, positive birth experience, initiation of breastfeeding in the early period, mother-infant bonding and transition to the role of motherhood .

İt will contribute positively to the health indicators of the country and reduce the cost, a scale and guide have been prepared within the scope of this thesis, with the foresight that pregnant women and health workers need training materials, and training with interactive and mobile communication tools in this direction. has been planned.It is expected that the training to be given in line with the developed guideline, and the empathic communication-based training given in the third trimester of pregnancy will help to increase the awareness of women's positive perception of birth.

With this study, it was aimed to determine the effect of empathic communication-based education on positive birth perception awareness.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older pregnancy

  * Speaks and understands Turkish
  * Able to read and write,
  * Having a single fetus,
  * Not having a risky pregnancy,
  * 32-36. in gestational week,
  * Pregnant women who do not have any disability diagnosed for normal delivery

Exclusion Criteria:

* Risky pregnant women
* Pregnant women with communication difficulties
* Pregnant women with mental deficiency

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2024-12-19 (Actual); Study Completion 2024-12-19 (Actual)

PRIMARY OUTCOMES:
Positive Birth Perception Awareness Scale | baseline
  Positive Birth Perception Awareness Scale (PDAFS): Focus group interviews will be held with 10-12 pregnant women for the scale to be developed. An item pool will be created from the themes and sub-areas obtained from the interviews. In addition, the factors affecting the awareness of positive birth perception of pregnant women were examined by examining the national and international literature, and a form will be prepared for the pilot study. The scale form, the literature study of the researchers and the findings of the focus group interviews will be re-evaluated and the pilot study form of the scale will be prepared. The pilot study form will be submitted to the expert opinion. The pilot form will be sent to 10-12 experts. By making arrangements in line with expert opinions, the question pool will be finalized before the application, and it will be transformed into a 5-point Likert scale model

SECONDARY OUTCOMES:
Wijma Birth Experience/Expectation Scale A (WBBSS-A) | baseline
  The scale consists of 33 items. The answers in the scale are in six-point Likert type numbered from 0 to 5. 0 is evaluated as "totally" and 5 as "not at all". The lowest score obtained from the scale is 0 and the highest score is 165. These; Those who have low level of fear of childbirth (WBLSS score ≤ 37), those who have moderate fear of childbirth (WBBSS-A score between 38-65).

CONTACTS AND LOCATIONS:
Overall Officials: Sultan ALAN, Principal Investigator — Çukuroava Universty; Emine AKSÜT AKÇAY, Principal Investigator — Kahramanmaraş Sütçü İmam Universty
Locations (1):
- Kahramanmaraş Sütçü İmam Universty, Kahramanmaraş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I do not approve of sharing ipd

REFERENCES:
- [Result] Karacam Z, Akyüz EÖ. Supportive care given in labor and the role of the midwife/nurse. FNJN 2011;19(1):45-5.
- [Result] Fullerton JT, Thompson JB, Severino R; International Confederation of Midwives. The International Confederation of Midwives essential competencies for basic midwifery practice. an update study: 2009-2010. Midwifery. 2011 Aug;27(4):399-408. doi: 10.1016/j.midw.2011.03.005. Epub 2011 May 20. PMID 21601321
- [Result] . Şenoğlu, A., & Karaçam, Z. Opinions and Needs of Birth Supporters on Participation in Birth. Dokuz Eylül University Faculty of Nursing Electronic Journal, 2019;12(4), 274-282.
- [Result] Lazzaretto E, Nespoli A, Fumagalli S, Colciago E, Perego S, Locatelli A. Intrapartum care quality indicators: a literature review. Minerva Ginecol. 2018 Jun;70(3):346-356. doi: 10.23736/S0026-4784.17.04177-6. Epub 2017 Nov 21. PMID 29161798
- [Result] Haapio S, Kaunonen M, Arffman M, Astedt-Kurki P. Effects of extended childbirth education by midwives on the childbirth fear of first-time mothers: an RCT. Scand J Caring Sci. 2017 Jun;31(2):293-301. doi: 10.1111/scs.12346. Epub 2016 Jul 21. PMID 27439382
- [Result] Toohill J, Callander E, Gamble J, Creedy DK, Fenwick J. A cost effectiveness analysis of midwife psycho-education for fearful pregnant women - a health system perspective for the antenatal period. BMC Pregnancy Childbirth. 2017 Jul 11;17(1):217. doi: 10.1186/s12884-017-1404-7. PMID 28693447
- [Result] Rouhe H, Salmela-Aro K, Toivanen R, Tokola M, Halmesmaki E, Ryding EL, Saisto T. Group psychoeducation with relaxation for severe fear of childbirth improves maternal adjustment and childbirth experience--a randomised controlled trial. J Psychosom Obstet Gynaecol. 2015;36(1):1-9. doi: 10.3109/0167482X.2014.980722. Epub 2014 Nov 24. PMID 25417935
- [Result] Lea J, Cruickshank M. Supporting new graduate nurses making the transition to rural nursing practice: views from experienced rural nurses. J Clin Nurs. 2015 Oct;24(19-20):2826-34. doi: 10.1111/jocn.12890. Epub 2015 Jul 14. PMID 26177875
- [Result] Oladapo OT, Tuncalp O, Bonet M, Lawrie TA, Portela A, Downe S, Gulmezoglu AM. WHO model of intrapartum care for a positive childbirth experience: transforming care of women and babies for improved health and wellbeing. BJOG. 2018 Jul;125(8):918-922. doi: 10.1111/1471-0528.15237. Epub 2018 May 15. No abstract available. PMID 29637727
- [Result] Ryding EL, Lukasse M, Parys AS, Wangel AM, Karro H, Kristjansdottir H, Schroll AM, Schei B; Bidens Group. Fear of childbirth and risk of cesarean delivery: a cohort study in six European countries. Birth. 2015 Mar;42(1):48-55. doi: 10.1111/birt.12147. PMID 25676793
- [Result] Navaee M, Abedian Z. Effect of role play education on primiparous women's fear of natural delivery and their decision on the mode of delivery. Iran J Nurs Midwifery Res. 2015 Jan-Feb;20(1):40-6. PMID 25709689
- [Result] Rouhe H, Salmela-Aro K, Toivanen R, Tokola M, Halmesmaki E, Saisto T. Obstetric outcome after intervention for severe fear of childbirth in nulliparous women - randomised trial. BJOG. 2013 Jan;120(1):75-84. doi: 10.1111/1471-0528.12011. Epub 2012 Nov 2. PMID 23121002
- [Result] Aktas S, Pasinlioglu T. The effect of empathy training given to midwives on the empathic communication skills of midwives and the birth satisfaction of mothers giving birth with the help of these midwives: A quasi-experimental study. J Eval Clin Pract. 2021 Aug;27(4):858-867. doi: 10.1111/jep.13523. Epub 2020 Dec 6. PMID 33283424
- [Result] Buchanan L, Anderson E, MBiostat HX, Phongsavan P, Rissel C, Wen LM. Sources of information and the use of mobile applications for health and parenting information during pregnancy: Implications for health promotion. Health Informatics J. 2021 Jul-Sep;27(3):14604582211043146. doi: 10.1177/14604582211043146. PMID 34569327
- [Result] Bogale B, Morkrid K, Abbas E, Abu Ward I, Anaya F, Ghanem B, Hijaz T, Isbeih M, Issawi S, A S Nazzal Z, E Qaddomi S, Froen JF. The effect of a digital targeted client communication intervention on pregnant women's worries and satisfaction with antenatal care in Palestine-A cluster randomized controlled trial. PLoS One. 2021 Apr 23;16(4):e0249713. doi: 10.1371/journal.pone.0249713. eCollection 2021. PMID 33891597
- [Result] Biaggi A, Conroy S, Pawlby S, Pariante CM. Identifying the women at risk of antenatal anxiety and depression: A systematic review. J Affect Disord. 2016 Feb;191:62-77. doi: 10.1016/j.jad.2015.11.014. Epub 2015 Nov 18. PMID 26650969
- [Result] Wijma K, Wijma B, Zar M. Psychometric aspects of the W-DEQ; a new questionnaire for the measurement of fear of childbirth. J Psychosom Obstet Gynaecol. 1998 Jun;19(2):84-97. doi: 10.3109/01674829809048501. PMID 9638601
- [Result] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Result] Dökmen Ü. Communication conflicts and empathy. 48th edition. Istanbul: Remzi Bookstore,2012.
- [Result] Gaskin IM. Ina May's Birth Preparation Guide. Erkök EE, Guler ZB (Transl). 1st edition. Istanbul: Sinek Eight Publishing House,2015.
- [Result] Cevik A, Alan S. Mental Health and Diseases for Midwives. Ed. Alan S. Pregnancy and Postpartum Period. Ankara; Academician Bookstore, 2019.